CLINICAL TRIAL: NCT05082051
Title: A 3-part, Phase 1a/1b, First-in-human, Randomized, Double-blind, Placebo-controlled Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of Oral CDX-7108 in Healthy Adult Subjects and to Evaluate Proof-of-concept Via Pharmacodynamics of a Single Dose of Oral CDX-7108 in Subjects with Exocrine Pancreatic Insufficiency
Brief Title: Oral CDX-7108 in Healthy Adults and EPI Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21.02.CLI
Record Dates: First submitted 2021-09-07; First posted 2021-10-18 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2023-04

CONDITIONS: Exocrine Pancreatic Insufficiency
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency | interventions — Medicare Part B; Medicare Part C

STUDY DESIGN:
Intervention Model Description: 3-part study Parts A and B are randomized, double-blind, placebo-controlled dose escalation parts to investigate the safety, tolerability, immunogenicity, and PK of CDX-7108 after single and multiple oral dose administration in healthy adult subjects. Part C is a randomized, double-blind, placebo-controlled, single-dose, 2-way crossover part to assess POC of CDX-7108 in terms of PD as well as its safety, tolerability, and immunogenicity in subjects with EPI.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CDX-7108 (Active Comparator): CDX-7108, an oral recombinant lipase. It is a modified version of a triacylglycerol lipase enzyme derived from the bacteria Bacillus thermoamylovans (btLIP) and produced by fermentation of recombinant Escherichia coli.7
  Interventions: Drug: Part A; Drug: Part B; Drug: Part C
- Placebo (Placebo Comparator): Excipients only
  Interventions: Drug: Part A; Drug: Part B; Drug: Part C

INTERVENTIONS:
Drug: Part A — Randomized, double-blind, placebo-controlled dose escalation part to investigate the safety, tolerability, immunogenicity, and PK of CDX-7108 after single oral dose administration in healthy adult subjects.
  Single-dose administration of CDX-7108 at the following anticipated dose levels. 10 000, 50 000, 150 000, 250 000, and 500 000 lipase units will be evaluated in 5 sequential cohorts of 6 subjects each.
  Other Names: Single Ascending Dose Study
Drug: Part B — Randomized, double-blind, placebo-controlled dose escalation parts to investigate the safety, tolerability, immunogenicity, and PK of CDX-7108 after multiple oral dose administration in healthy adult subjects.
  It will evaluate multiple dose administration of CDX-7108 at an appropriate low (50 000 lipase units), mid (150 000 lipase units), and high dose (250 000 lipase units) 4 times a day (QID) for 6 consecutive days in 3 sequential cohorts of 6 subjects each.
  Other Names: Multiple Ascending Dose Study
Drug: Part C — Randomized, double-blind, placebo-controlled, single-dose, 2-way crossover part to assess POC of CDX-7108 in terms of PD as well as its safety, tolerability, and immunogenicity in subjects with EPI.
  Approximately 10 subjects with severe EPI from partial/total pancreatectomy or chronic pancreatitis will be enrolled. It is anticipated that Part C (POC study) will commence after completion of the third single-dose cohort from Part A (SAD study) and following SRC review of the data from this cohort.
  Other Names: Proof-of-Concept Study

SUMMARY:
Phase 1a/1b single and multiple ascending dose study of oral CDX-7108 in healthy adult subjects and a single dose proof-of-concept study of oral CDX-7108 in subjects with exocrine pancreatic insufficiency.

No clinical studies have yet been performed with CDX-7108 and its effects in humans are unknown. This is the first-in-human (FIH) study of CDX-7108, which aims to assess the safety, tolerability, pharmacokinetics (PK) of escalating single and multiple oral doses of CDX-7108 in healthy adult subjects and to evaluate the pharmacodynamics of a single dose of oral CDX-7108 in a proof-of-concept (POC) study in subjects with exocrine pancreatic insufficiency (EPI).

DETAILED DESCRIPTION:
This is an integrated 3-part study to investigate the safety, tolerability, PK, and PD of CDX-7108. The Parts A and B are randomized, double-blind, placebo-controlled dose escalation parts to investigate the safety, tolerability, immunogenicity, and PK of CDX-7108 after single and multiple oral dose administration in healthy adult subjects. Part C is a randomized, double-blind, placebo-controlled, single-dose, 2-way crossover part to assess POC of CDX-7108 in terms of PD as well as its safety, tolerability, and immunogenicity in subjects with EPI. The study will commence with Part A (single ascending dose [SAD] study) and will progress to Part B (multiple ascending dose [MAD] study), and Part C (POC study)

ELIGIBILITY:
Inclusion Criteria:

All subjects:

1. Capable of giving signed informed consent prior to initiation of any protocol-specific procedures, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Body mass index (BMI) between 18.0 and 30.0 kg/m2.
3. Nonsterilized male subjects are eligible to participate if they agree to ONE of the following starting at Screening and continuing throughout the clinical study period, and for 90 days after IP administration:

   1. Must agree to stay abstinent (where abstinence is the preferred and usual lifestyle of the subject), OR
   2. Male subjects with a female partner of childbearing potential must agree to use highly effective contraception consisting of 2 forms of birth control.
   3. Male subjects with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or use a male condom during each episode of penile penetration.
   4. These requirements do not apply to subjects in a same sex relationship.
4. Male subjects must agree not to donate sperm starting at Screening and continuing throughout the clinical study period, and for 90 days after IP administration.
5. Female subjects of childbearing potential are eligible to participate if they meet the following criteria:

   1. Must agree not to become pregnant during the clinical study period and for 30 days after IP administration.
   2. Must have a negative serum pregnancy test at Screening and Day -1.
   3. If heterosexually active, must agree to consistently use a form of highly effective birth control, in combination with a barrier method (as defined in Appendix 3) starting at Screening (signing the ICF) and continuing throughout the clinical study period, and for 30 days after IP administration, OR
   4. Must agree to stay abstinent (where abstinence is the preferred and usual lifestyle of the subject), starting at Screening (signing the ICF) and continuing throughout the clinical study period, and for 30 days after IP administration.
   5. These requirements do not apply to subjects in a same sex relationship.
6. Female subjects of non-childbearing potential are eligible to participate if 1 of the following conditions apply:

   1. Must have a confirmed clinical history of sterility (documented hysterectomy, bilateral salpingectomy, or bilateral oophorectomy, as confirmed by review of the subject's medical records, medical examination, or medical history interview)
   2. Must be postmenopausal as defined as: amenorrhea for at least 1 year prior to Screening and a laboratory confirmed serum follicle-stimulating hormone (FSH) level ≥40 mIU/mL. Female subjects on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use 1 of the non-estrogen hormonal highly effective contraception methods (Appendix 3) from Screening (signing the ICF) until at and continuing throughout the clinical study period, and for 30 days after IP administration if they wish to continue their HRT during the study.
7. Female subjects must agree not to donate ova starting at Screening (signing the ICF) and continuing throughout the clinical study period, and for 30 days after IP administration.
8. Subject agrees not to participate in another interventional study while participating in the present clinical study.

   Parts A (Single Ascending Dose Study) and B (Multiple Ascending Dose Study)
9. Healthy male and female, non-smoking, subjects between the ages of 18 and 55 years, inclusive, at the time of Screening. In each cohort, at least 2 male subjects and 2 female subjects should be enrolled.
10. Appropriate general health, as determined by an experienced physician based on a medical evaluation including detailed medical history, clinical laboratory tests, vital signs, 12-lead ECG, and full physical examination (and neurological assessment).

    Part C (Proof-of-Concept Study)
11. Male and female subjects between the ages of 18 and 75 years (inclusive) who have undergone total or partial pancreatectomy or have an established diagnosis of CP, as confirmed by fecal pancreatic elastase-1 <100 μg/g in formed stools within 12 months of the Screening visit.
12. Subjects with clinically well controlled EPI under the regular use of PERT (remission or adequate improvement of steatorrhea on PERT), as determined by an experienced physician based on a medical evaluation including detailed medical history, clinical laboratory tests, vital signs, 12-lead ECG, and full physical examination (and neurological assessment).
13. 150min percentage 13CO2 excretion rate <4.4% dose/h using the Pancreo-Lip breath test at Screening.

Exclusion Criteria:

All subjects

1. Female subject who has been pregnant within the 6 months prior to Screening or breastfeeding within the 3 months prior to Screening.
2. Treatment with any antiplatelet and/or anticoagulant medication, except low-dose aspirin.
3. Evidence or history of specific food intolerance. Examples include gluten intolerance, lactose intolerance, or dairy food intolerance or any food/ingredient included in the standard breakfast provided at the study site.
4. A positive result, on Screening, for serum hepatitis B surface antigen, hepatitis A virus antibodies, hepatitis C virus antibodies or antibodies to human immunodeficiency virus type 1 and/or type 2.
5. Known active infection with COVID-19, or a suspected infection with severe acute respiratory syndrome coronavirus-2 [SARS-CoV-2]).
6. Chronic alcoholic intoxication that would preclude compliance with the study procedures.
7. Habitual use of nicotine products or smoking within 3 months (>10 cigarettes per day) prior to Screening, and/or unwilling to refrain from smoking during the confinement period. Nicotine replacement therapy is allowed during the study.
8. Drug addiction that would preclude participation and compliance with study procedures.
9. Subject has a pulse rate <40 or >100 bpm; mean systolic blood pressure (SBP) >150 mmHg; mean diastolic blood pressure (DBP) >95 mmHg at Screening. Repeat measurements are allowed at the discretion of the Investigator.
10. Subject has any clinically significant abnormalities at Screening in rhythm, conduction or morphology of the resting ECG and any clinically significant abnormalities in the 12-lead ECG, as considered by the Investigator, that may interfere with the interpretation of QTc interval changes including abnormal ST-T wave morphology.
11. Subject has prolonged QTcF >450 msec for male subjects or >470 msec for female subjects or a family history of prolonged QT syndrome, at Screening.
12. Plasma donation within the 14 days prior to the first dose of IP or any whole blood donation/significant blood loss >500 mL during the 3 months prior to the first dose of IP.
13. Treatment with any investigational drug or device/treatment within the 30 days or 5 half-lives of the drug (whichever is longer) prior to the administration of IP.
14. Known allergy or adverse reaction history to any component of the CDX-7108 oral dose formulation.

    Part A (Single Ascending Dose Study) and Part B (Multiple Ascending Dose Study)
15. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies and childhood asthma) at time of Screening or IP administration, that in the opinion of the Investigator may put the subject at greater safety risk, influence response to study drug, or interfere with study assessments.
16. Current or chronic history of GI disorders or conditions interfering with normal GI anatomy or function. Examples include GI bypass surgery, partial or total gastrectomy, gastric band surgery, major (>1 m) small bowel resection, vagotomy, malabsorption, Crohn's disease, ulcerative colitis, irritable bowel syndrome, celiac sprue, and small intestinal bacterial overgrowth.
17. A positive Screening test for use of drugs (amphetamines, cocaine, marijuana, opiates, barbiturates, benzodiazepines, methadone, and methamphetamines) and alcohol (breath test). However, there is the option to re-screen once during the Screening period at the discretion of the Investigator or delegate in the case of a positive result at Screening for a prescribed medication, eg, codeine.
18. Subject has any clinically significant abnormalities in hematology, coagulation, clinical chemistry, or urinalysis at Screening as judged by the Investigator, including aspartate aminotransferase (AST) or ALT >1.5 times above the ULN. Repeat measurements are allowed at the discretion of the Investigator.
19. Use of any prescribed or nonprescribed medication in the 2 weeks preceding the first dose of IP. EXCEPTION: Subjects who have received approved vaccines (including approved COVID-19 vaccines) may be allowed if these vaccines are taken no less than 72 hours prior to the IP dose at the discretion of the Investigator.

    Part C (Proof-of-Concept Study)
20. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies and childhood asthma) at time of Screening or IP administration, that in the opinion of the Investigator may put the subject at greater safety risk, influence response to study drug, or interfere with study assessments. NOTE: Subjects with treated diabetes secondary to CP or pancreatectomy are allowed.
21. Subject has any clinically significant abnormalities in hematology, coagulation, clinical chemistry, or urinalysis at Screening as judged by the Investigator, including AST or ALT >1.5 times above the ULN, or cholesterol or triglycerides >400 mg/dL. Repeat measurements are allowed at the discretion of the Investigator.
22. Current or chronic history of GI disorders or conditions interfering with normal GI anatomy or motility, with the exception of pancreatic insufficiency due to pancreatectomy, including pancreaticoduodenectomy, or CP
23. Use of any prescribed or nonprescribed medication potentially interfering with gastric pH, intestinal motility, or fat absorption, including herbal and dietary supplements and antacids; these medications shall be stopped for a minimum of 5 times their half-life before IP administration if, in the opinion of the Investigator, this does not represent a risk for the subject's wellbeing. EXCEPTIONS:

    Histamine H2 receptor antagonists, PPI, insulin, analgesics, and chronic pain medications.

    Oral contraceptives, paracetamol, or multivitamins. Subjects who have received approved vaccines (including approved COVID-19 vaccines) may be allowed if these vaccines are taken no less than 72 hours prior to the IP dose at the discretion of the Investigator.
24. Use of antibiotics within 8 days before the Pancreo-Lip breath test at Screening or Day 1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Adverse events | Up to 9 weeks
  Number and severity of adverse events
Changes in haematology from baseline | Up to 5 weeks
  Number of participants with changes in haematology measurements (erythrocyte count, thrombocyte count, haemoglobin, haematocrit, mean cell hemoglobin concertation) using immunoassays.
Changes in coagulation tests from baseline | Up to 5 weeks
  Number of participants with changes in coagulation factors (INR, prothrombin time, fibrogen, red blood cell indices and leukocyte count) using immunoassays.
Changes in clinical chemistry from baseline | Up to 5 weeks
  Number of participants with changes in clinical chemistry (bicarbonate, albumin, total protein, blood glucose, sodium, potassium, phosphate, calcium, urea creatine, chloride, creatine kinase, urate, AST, ALT, ALP, GGT, triglycerides, total cholesterol, lactate dehydrogenase, c-reactive protein, total bilirubin) using immunoassays.
Changes in urinalysis from baseline | Up to 5 weeks
  Number of participants with changes in leucocyte esterase, protein, urobilinogen, ketones, bilirubin, microscopy, blood, pH, nitrate, specific gravity, urobilinogen and glucose) using immunoassays.
Changes in Systolic Blood Pressure from baseline | Up to 5 weeks
  Changes in Systolic Blood Pressure from baseline
Changes in Diastolic Blood Pressure from baseline | Up to 5 weeks
  Changes in Diastolic Blood Pressure from baseline
Changes in Pulse Rate vital signs from baseline | Up to 5 weeks
  Changes in pulse rate from baseline
Changes in Respiratory Rate vital signs from baseline | Up to 5 weeks
  Changes in respiratory rate from baseline
Changes in Body Temperature vital signs from baseline | Up to 5 weeks
  Changes in body temperature from baseline
Changes in 12-lead electrocardiogram (ECG) Heart Rate from baseline | Up to 5 weeks
  Changes in ECG Heart rate from baseline
Changes in 12-lead electrocardiogram (ECG) PR Interval from baseline | Up to 5 weeks
  Changes in ECG PR interval from baseline
Changes in 12-lead electrocardiogram (ECG) QRS duration from baseline | Up to 5 weeks
  Changes in electrocardiogram QRS duration interval from baseline
Changes in 12-lead electrocardiogram (ECG) QT Interval from baseline | Up to 5 weeks
  Changes in ECG QT interval from baseline
Changes in 12-lead electrocardiogram (ECG) QTcF Interval from baseline | Up to 5 weeks
  Changes in ECG QTcF interval from baseline
Changes in physical examination from baseline: Head | Up to 5 weeks
  Changes in general appearance of the head from baseline
Changes in physical examination from baseline: Ears | Up to 5 weeks
  Changes in general appearance of the ears from baseline
Changes in physical examination from baseline: Eyes | Up to 5 weeks
  Changes in general appearance of the eyes from baseline
Changes in physical examination from baseline: Nose | Up to 5 weeks
  Changes in general appearance of the nose from baseline
Changes in physical examination from baseline: Throat | Up to 5 weeks
  Changes in general appearance of the throat from baseline
Changes in physical examination from baseline: Neck | Up to 5 weeks
  Changes in general appearance of the neck (including thyroid) from baseline
Changes in physical examination from baseline: General Appearance | Up to 5 weeks
  Changes in general appearance of the skin from baseline
Changes in physical examination from baseline: Cardiovascular system | Up to 5 weeks
  Changes in cardiovascular system from baseline
Changes in physical examination from baseline: Respiratory system | Up to 5 weeks
  Changes in respiratory system from baseline
Changes in physical examination from baseline: GI system | Up to 5 weeks
  Changes in GI system from baseline
Changes in physical examination from baseline: Musculoskeletal system | Up to 5 weeks
  Changes in musculoskeletal system from baseline
Changes in physical examination from baseline: Lymph nodes | Up to 5 weeks
  Changes in lymph nodes from baseline
Changes in physical examination from baseline: Nervous system | Up to 5 weeks
  Changes in nervous system from baseline

SECONDARY OUTCOMES:
Concentration-time profile of CDX-7108 | Up to 7 days
  Serum concentration-time profile of CDX-7108
Lipase activity | Day 1
  Serum Lipase activity
CO2 excretion rate | Up to 43 days
  CO2 excretion rate (% dose/h),

OTHER OUTCOMES:
Immunogenicity Assessment | Up to 5 weeks
  Serum anti-CDX-7108 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Chris Wynne, Principal Investigator — New Zealand Clinical Research; John Windsor, Principal Investigator — New Zealand Clinical Research; Nam Nguyen, Principal Investigator — CMAX Clinical Research; Richard Stubbs, Principal Investigator — P3 Research
Locations (4):
- CMAX Clinical Research, Adelaide, New South Wales, Australia
- New Zealand (3):
  - New Zealand Clinical Research, Auckland, North Island
  - New Zealand Clinical Research, Christchurch, South Island
  - P3 Research, Lower Hutt, Wellington Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forsmark Chris E. Chronic pancreatitis In: Sleisenger M, Fordtran J, Feldman M, Brandt L, and Friedman L. eds. Sleisenger & Fordtran's Gastrointestinal and liver disease. 10th ed Philadelphia, PA: Saunders-Elsevier; 2016:1020.
- [Background] Shandro BM, Nagarajah R, Poullis A. Challenges in the management of pancreatic exocrine insufficiency. World J Gastrointest Pharmacol Ther. 2018 Oct 25;9(5):39-46. doi: 10.4292/wjgpt.v9.i5.39. PMID 30397535
- [Background] ASGE Standards of Practice Committee; Chandrasekhara V, Chathadi KV, Acosta RD, Decker GA, Early DS, Eloubeidi MA, Evans JA, Faulx AL, Fanelli RD, Fisher DA, Foley K, Fonkalsrud L, Hwang JH, Jue TL, Khashab MA, Lightdale JR, Muthusamy VR, Pasha SF, Saltzman JR, Sharaf R, Shaukat A, Shergill AK, Wang A, Cash BD, DeWitt JM. The role of endoscopy in benign pancreatic disease. Gastrointest Endosc. 2015 Aug;82(2):203-14. doi: 10.1016/j.gie.2015.04.022. Epub 2015 Jun 12. No abstract available. PMID 26077456
- [Background] Saito T, Hirano K, Isayama H, Nakai Y, Saito K, Umefune G, Akiyama D, Watanabe T, Takagi K, Hamada T, Takahara N, Uchino R, Mizuno S, Kogure H, Matsubara S, Yamamoto N, Tada M, Koike K. The Role of Pancreatic Enzyme Replacement Therapy in Unresectable Pancreatic Cancer: A Prospective Cohort Study. Pancreas. 2017 Mar;46(3):341-346. doi: 10.1097/MPA.0000000000000767. PMID 28099252
- [Background] Imrie CW, Connett G, Hall RI, Charnley RM. Review article: enzyme supplementation in cystic fibrosis, chronic pancreatitis, pancreatic and periampullary cancer. Aliment Pharmacol Ther. 2010 Nov;32 Suppl 1:1-25. doi: 10.1111/j.1365-2036.2010.04437.x. PMID 21054452
- [Background] Keller J, Layer P. Human pancreatic exocrine response to nutrients in health and disease. Gut. 2005 Jul;54 Suppl 6(Suppl 6):vi1-28. doi: 10.1136/gut.2005.065946. No abstract available. PMID 15951527
- [Background] Investigator's Brochure for CDX-7108. Edition 1.0, Release Date 31 March 2021.
- [Background] CREON®. The United States Prescribing Information. Available at: https://www.accessdata.fda.gov/drugsatfda_docs/label/2009/020725s000lbl.pdf. Accessed on: 23 March 2021.
- [Background] Food and Drug Administration. Guidance for industry: estimating the maximum safe starting dose in initial clinical trials for therapeutics in adult healthy volunteers. Center for Drug Evaluation and Research (CDER). 2005.
- [Background] Food and Drug Administration. Guidance for industry drug-induced liver injury: premarketing clinical evaluation. CDER. 2009.
- [Background] Loser C, Brauer C, Aygen S, Hennemann O, Folsch UR. Comparative clinical evaluation of the 13C-mixed triglyceride breath test as an indirect pancreatic function test. Scand J Gastroenterol. 1998 Mar;33(3):327-34. doi: 10.1080/00365529850170946. PMID 9548629
- [Background] Aygen S, inventor; Infai Institut fur Biomedizinische Analytik und NMR Imaging GmbH, assignee. Method for measuring pancreatic metabolism. International Patent, WO2004043498. 27 May 2004.
- [Background] Aygen S, inventor; Infai Institut fur Biomedizinische Analytik und NMR Imaging GmbH, assignee. Method for measuring pancreatic metabolism. European Patent, EP1560603. 07 March 2007.
- [Background] Aygen S, inventor; Infai Institut fur Biomedizinische Analytik und NMR Imaging GmbH, assignee. Method for measuring pancreatic metabolism. United States patent US 7762957. 27 July 2010.
- [Background] James LP, Letzig L, Simpson PM, Capparelli E, Roberts DW, Hinson JA, Davern TJ, Lee WM. Pharmacokinetics of acetaminophen-protein adducts in adults with acetaminophen overdose and acute liver failure. Drug Metab Dispos. 2009 Aug;37(8):1779-84. doi: 10.1124/dmd.108.026195. Epub 2009 May 13. PMID 19439490